CLINICAL TRIAL: NCT00726674
Title: Lantus for Diabetic Patients Treated in Clalit Outpatient Clinics
Brief Title: Basal Insulin for Type 2 Diabetes Patients Treated in Outpatient Clalit Clinics
Acronym: Lapas II
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: LANTU_L_04137
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes HbA1C
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Treatment of diabetes mellitus type II with basal insulin, for patients treated in Clalit outpatient clinics that are not adequately controlled with current treatment.

DETAILED DESCRIPTION:
Patients with diabetes treated in outpatient clinics will be recruited by their primary care physician. Recruitment period will be 3 months per center and each patient will be followed for 7 months Diabetes specialists will be responsible for 50-65 primary care physicians. The specialists will advise and direct the primary care physician through the whole study period.

The study protocol includes patients treated with different types of non short- acting insulin. Insulin Lantus (including dose) will be started by the primary physician, if needed after consulting the Diabetes Specialist. The treatment should follow the study protocol.

Patients will have 3 pre-scheduled visits in their clinic: 1. At the beginning of study. 2. After 3 months. 3. At study end (after 6 month). An additional telephone contact will take place 1 month after last visit. to evaluate adherence to therapy Data collecting: Data including HbA1c, FPG,current diabetic treatment, dose of insulin Lantus, and relevant additional diseases\complaints will be collected at each visit. Additional information as demographic data, medical history will be collected at beginning of study.

Safety: Hypoglycaemic episodes will be recorded

ELIGIBILITY:
Inclusion Criteria:

1. Type II Diabetic patients
2. HbA1c >8.0% (result from preceding 4 months)
3. Written informed consent
4. Life expectancy of at least 1 year.
5. Patients' agree to discontinue current long acting insulin (if applicable).
6. Patients who according to their GP are eligible to the study.

Exclusion Criteria:

1. Type I diabetes
2. Pregnancy and\or lactation.
3. Allergy to basal insulin
4. Patients suffering from a disease that requires repeated hospitalizations E.g.: severe CHF, sever renal failure, active malignancy.
5. Patients who are not able to give consent.
6. Patients face difficulties in mobility and/or verbal communication with the treating physician.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type II diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 1229 (Actual)
Dates: Start 2008-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Decrease in HbA1c level | 6 months

SECONDARY OUTCOMES:
Safety measures | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Nurit Tweezer-Zaks, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Netanya, Israel